CLINICAL TRIAL: NCT05414565
Title: Clinical and Functional Performance of Acrysof IQ Vivity Versus Aspheric Monofocal IOLs
Brief Title: Post-Market Study of Alcon Intraocular Lenses
Status: Completed | Type: Observational
Sponsor: Alcon Research (Industry)
Collaborators: Queensland University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: A04429
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Visual Acuity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vivity IOL: Subjects previously implanted with Vivity or Vivity toric IOL
  Interventions: Device: Vivity IOL
- Aspheric Monofocal IOL: Subjects previously implanted with an aspheric monofocal or monofocal toric IOL
  Interventions: Device: Aspheric monofocal IOL

INTERVENTIONS:
Device: Vivity IOL — Commercially available extended vision IOL
  Other Names: Acrysof IQ Vivity or Vivity toric IOL
  Groups: Vivity IOL
Device: Aspheric monofocal IOL — Commercially available aspheric IOL
  Other Names: Acrysof IQ monofocal or monofocal toric IOL; Clareon monofocal or monofocal toric IOL
  Groups: Aspheric Monofocal IOL

SUMMARY:
The purpose of the study is to evaluate clinical and functional performance in real-world conditions in participants who have been implanted with Acrysof IQ Vivity (Extended Vision) IOLs compared with Alcon Aspheric Monofocal IOLs.

DETAILED DESCRIPTION:
This observational study will enroll subjects who have been implanted with an Alcon aspheric monofocal or monofocal toric IOL no less than 4 months prior to study procedures. This study will be conducted in Australia.

ELIGIBILITY:
Key Inclusion Criteria:

* In good general health at the screening visit;
* Implanted in both eyes at least 4 months ago with either Vivity/Vivity toric IOL or an Alcon aspheric monofocal/monofocal toric IOL (Acrysof IQ/Clareon);
* Best Corrected Distance Visual Acuity (BCDVA) of 20/25 or better with both eyes together;
* BCDVA of 20/40 or better in each eye;

Key Exclusion Criteria:

* Clinically significant Posterior Capsular Opacity (PCO) as assessed via slit-lamp exam per investigator opinion;
* History of ocular surgery other than cataract surgery and Nd:YAG laser surgery;
* History of amblyopia.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from ophthalmology practices who implant the Alcon Vivity and Alcon aspheric monofocal IOLs.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Binocular photopic best-corrected distance visual acuity (BCDVA) | At least 4 months post-operative
  Visual acuity will be measured using a standard visual acuity chart at a distance of 4 meters under photopic (well-lit) conditions and reported in logarithm Minimum Angle of Resolution (logMAR) units. Visual acuity will be measured binocularly (both eyes together).

CONTACTS AND LOCATIONS:
Overall Officials: Director of Clinical Projects, Surgical, Study Director — Alcon Research, LLC
Locations (1):
- School of Optometry and Vision Science, Queensland University of Technology, Kelvin Grove, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No